CLINICAL TRIAL: NCT01469065
Title: A 2-week, Phase 1, Placebo-Controlled, Parallel Group Trial To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Multiple Oral Doses Of PF-04991532 Given As Monotherapy To Adult Patients With Type 2 Diabetes Mellitus
Brief Title: A 2-week Trial Of PF-04991532 In Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B2611005
Record Dates: First submitted 2011-10-25; First posted 2011-11-10 (Estimated); Results first posted 2013-08-29 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: inpatient; diabetes; phase 1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — 6-(3-cyclopentyl-2-(4-(trifluoromethyl)-1H-imidazol-1-yl)propanamido)nicotinic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04991532 (Experimental): PF-04991532 experimental study medication
  Interventions: Drug: PF-04991532; Drug: PF-0499132
- Placebo (Placebo Comparator): PF-04991532 Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04991532 — Oral administration of PF-04991532; 25 mg given twice a day (BID) for 14 days
  Arms: PF-04991532
Drug: PF-04991532 — Oral administration of PF-04991532; 75 mg given twice a day (BID) for 14 days
  Arms: PF-04991532
Drug: PF-04991532 — Oral administration of PF-04991532; 150 mg given twice a day (BID) for 14 days
  Arms: PF-04991532
Drug: PF-0499132 — Oral administration of PF-04991532; 300 mg given twice a day (BID) for 14 days
  Arms: PF-04991532
Drug: Placebo — Oral administration of PF-04991532 Matching Placebo; given twice a day (BID) for 14 days
  Arms: Placebo

SUMMARY:
This will be a 2-week oral dose study of PF 04991532, performed in patients with type 2 diabetes. Safety, pharmacokinetics (how the drug is distributed in the body), and pharmacodynamics (how the drug works in the body) will be studied. Patients may be asked to wash off their diabetes medication for 4-6 prior to study drug administration, and they will remain in the clinical research unit for a total of 20 days for baseline tests, 2 weeks of dosing, and some follow up tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus who are taking either no medication for the treatment of diabetes (diet/exercise therapy only), or who are taking only a single oral anti-diabetic drug (OAD) that can be temporarily discontinued for approximately 8-10 weeks. For those taking a single OAD, treatment should be stable, where this is defined as no change in the treatment, including dose, over the past 3 months prior to Screening. OAD medications that are acceptable to be discontinued include: a sulfonylurea (SU), a meglitinide, a biguanide (eg, metformin), a dipeptidyl peptidase 4 inhibitor (DPP-4i), or an alpha glucosidase inhibitor.
* Body Mass Index (BMI) of 18.5 to 45.0 kg/m2; and a total body weight >50 kg (110 lbs).
* HbA1c >/=7% and </=10% if the patient is on diet/exercise therapy only and does not require any OAD discontinuation. HbA1c >/=6.5% and </=9% if the patient requires to be washed off an OAD.

Exclusion Criteria:

* Evidence or history of diabetic complications with significant end organ damage.
* History of stroke or transient ischemic attack.
* History of myocardial infarction.
* History of coronary artery bypass graft or stent implantation.
* Clinically significant peripheral vascular disease.
* Any history or clinical evidence of congestive heart failure, NYHA Classes II IV.
* Current history of angina/unstable angina.
* One or more episodes of hypoglycemia within the last 3 months, or two or more episodes of hypoglycemia within the last 6 months.
* A positive urine drug screen.
* Use of tobacco or nicotine-containing products in excess of the equivalent of 10 cigarettes per day.
* Blood pressure >/=160 mm Hg (systolic) or >/=100 mm Hg (diastolic), following at least 5 minutes of rest.
* Pregnant or nursing females; females of childbearing potential.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (2):
  - Pfizer Investigational Site, Chula Vista, California
  - Pfizer Investigational Site, Miami, Florida
- Pfizer Investigational Site, Hachioji-shi, Tokyo, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2611005&StudyName=A%202-week%20Trial%20Of%20PF-04991532%20In%20Patients%20With%20Type%202%20Diabetes

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: PF-04991532 matching placebo orally twice daily for 2 weeks.
- PF-04991532 25 mg: PF-04991532 25 milligram (mg) tablet orally twice daily for 2 weeks.
- PF-04991532 75 mg: PF-04991532 75 mg tablet orally twice daily for 2 weeks.
- PF-04991532 150 mg: PF-04991532 150 mg tablet orally twice daily for 2 weeks.
- PF-04991532 300 mg: PF-04991532 300 mg tablet orally twice daily for 2 weeks.
Period: Overall Study
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Started | 16 | 17 | 16 | 16 | 17
Completed | 16 | 16 | 16 | 16 | 16
Not Completed | 0 | 1 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg | Total
Number analyzed (Participants) | 16 | 17 | 16 | 16 | 17 | 82
Age Continuous [Mean (Standard Deviation); unit: years] | 59.2 (8.2) | 56.4 (9.0) | 57.4 (10.7) | 57.0 (9.4) | 56.1 (8.0) | 57.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 2 | 5 | 20
  Male | 12 | 13 | 11 | 14 | 12 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Day -1) in Mean Daily Glucose at Day 14
Description: Mean daily glucose (MDG) was calculated based on the mean of 8 glucose measurements at pre-specified time points throughout the day on Day -1 and Day 14.
Time Frame: Baseline: hours -46, -44, -42, -40, -38, -36, -33, -and -30 on Day -1 (Day 1 morning dose was hour 0); Day 14: 2, 4, 6, 8, 10, 12, 15, and 18 hours after Day 14 morning dose
Population: The pharmacodynamic analysis population was defined as all randomized participants who received at least 1 dose of study medication (PF-04991532 or placebo) and had at least 1 of the pharmacodynamic parameters of interest.
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
milligram/deciliter (mg/dL)
  Baseline (Day -1) | 228.67 (36.26) | 233.20 (41.01) | 219.13 (38.16) | 229.92 (52.93) | 218.20 (53.01)
  Change from Baseline (Day 14) | 24.98 (40.48) | -17.55 (25.40) | -3.67 (33.79) | -9.73 (21.52) | -29.23 (32.80)
Statistical Analysis 1: Comparison: Placebo vs PF-04991532 25 mg; Test-to-Reference ratio and 90% confidence interval (CI) were based on adjusted geometric mean. Natural log-transformed change from baseline in MDG (Day 14) was analyzed using ANCOVA with country and treatment as fixed effect and log-transformed baseline as covariate. Placebo is the reference; the active drug group is the test. Formal statistical inference was not performed thus p value was not reported; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 84.87, 90% CI 2-sided [78.16 to 92.15]
Statistical Analysis 2: Comparison: Placebo vs PF-04991532 75 mg; Test-to-Reference ratio and 90% confidence interval (CI) were based on adjusted geometric mean. Natural log-transformed change from baseline in MDG (Day 14) was analyzed using ANCOVA with country and treatment as fixed effect and log-transformed baseline as covariate. Placebo is the reference; the active drug group is the test; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 89.80, 90% CI 2-sided [82.69 to 97.53]
Statistical Analysis 3: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 87.15, 90% CI 2-sided [80.27 to 94.63]
Statistical Analysis 4: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 78.28, 90% CI 2-sided [72.06 to 85.03]

2. Secondary Outcome: Area Under the Curve From Time Zero to 24 Hours Postdose (AUC24) of PF-04991532
Description: Area under the plasma concentration versus time curve (AUC) from time zero to 24 hours post morning dose
Time Frame: 0 (before morning dose), 0.5, 1, 2, 3, 4, 6, 10, 10.5, 11, 12, 13, 15, 18, and 24 hours after morning dose on Day 1 and Day 14
Population: The pharmacokinetic parameter analysis population was defined as all randomized participants treated with PF-04991532 who had at least 1 of the pharmacokinetic parameters of interest; "n" is the number of participants analyzed for each day.
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 16 | 16 | 16 | 17
nanogram*hour/milliliter (ng*hr/mL)
  Day 1 (n=16, 16, 16, 17) | 441.6 (172.3) | 1745 (757.1) | 3899 (1549) | 6943 (3053)
  Day 14 (n=16, 16, 16, 16) | 487.4 (227.1) | 1892 (930.1) | 3870 (1369) | 7531 (3084)

3. Secondary Outcome: Area Under the Curve From Time Zero to 10 Hours Postdose (AUC10) of PF-04991532
Description: Area under the plasma concentration versus time curve (AUC) from time zero to 10 hours post morning dose.
Time Frame: 0 (before morning dose), 0.5, 1, 2, 3, 4, 6, and 10 hours after morning dose on Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 16 | 16 | 16 | 17
ng*hr/mL
  Day 1 (n=16, 16, 16, 17) | 372.1 (146.7) | 1447 (749.3) | 3329 (1153) | 5661 (2595)
  Day 14 (n=16, 16, 16, 16) | 384.7 (181.9) | 1508 (920.7) | 2882 (1128) | 5551 (2633)

4. Secondary Outcome: Maximum Observed Plasma Concentration of PF-04991532 After Morning Dose Administration (Cmax(AM))
Time Frame: 0 (before morning dose), 0.5, 1, 2, 3, 4, 6, and 10 hours after morning
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 17 | 16 | 16 | 17
ng/mL
  Day 1 (n=17, 16, 16, 17) | 137.7 (57.36) | 486.6 (363.7) | 1285 (585.8) | 1951 (1106)
  Day 14 (n=16, 16, 16, 16) | 148.2 (74.23) | 469.8 (495.3) | 902.4 (489.1) | 1639 (917.8)

5. Secondary Outcome: Maximum Observed Plasma Concentration of PF-04991532 After Evening Dose Administration (Cmax(PM))
Time Frame: 10 (before evening dose), 10.5, 11, 12, 13, 15, 18, and 24 hours after morning dose on Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 16 | 16 | 16 | 17
ng/mL
  Day 1 (n=16, 16, 16, 17) | 97.10 (67.45) | 336.0 (219.7) | 932.0 (387.7) | 1645 (1132)
  Day 14 (n=16, 16,16, 16) | 89.99 (46.05) | 360.7 (288.8) | 772.4 (310.8) | 1687 (914.9)

6. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) of PF-04991532
Time Frame: Day 14
Population: The pharmacokinetic parameter analysis population was defined as all randomized participants treated with PF-04991532 who had at least 1 of the pharmacokinetic parameters of interest.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng/mL | 0.1691 (1.373) | 5.249 (3.112) | 11.32 (8.126) | 21.15 (12.73)

7. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-04991532 After Morning Dose Administration (Tmax(AM))
Time Frame: 0 (predose), 0.5, 1, 2, 3, 4, 6, and 10 hours after morning dose on Day 1 and Day 14
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 17 | 16 | 16 | 17
hour
  Day 1 (n=17, 16, 16, 17) | 1.00 [0.500 to 1.95] | 1.00 [0.500 to 6.00] | 1.83 [1.00 to 1.95] | 1.00 [0.500 to 3.00]
  Day 14 (n=16, 16, 16, 16) | 1.00 [0.500 to 1.95] | 1.00 [0.500 to 6.00] | 1.83 [0.500 to 6.00] | 1.45 [1.00 to 6.00]

8. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-04991532 After Evening Dose Administration (Tmax(PM))
Description: Time was computed as post morning dose.
Time Frame: 10 (before evening dose), 10.5, 11, 12, 13, 15, 18, and 24 hours after morning dose on Day 1 and Day 14
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 16 | 16 | 16 | 17
hour
  Day 1 (n=16, 16, 16, 17) | 11.0 [11 to 15] | 11.0 [11 to 15] | 11.0 [11 to 12] | 11.0 [11 to 13]
  Day 14 (n=16, 16, 16, 16) | 11.0 [11 to 15] | 11.0 [11 to 15] | 11.0 [11 to 18] | 11.0 [11 to 18]

9. Secondary Outcome: Apparent Oral Clearance (CL/F) of PF-04991532
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Day 1 and Day 14: 0 (before morning dose), 0.5, 1, 2, 3, 4, 6, 10 (before evening dose), 10.5, 11, 12, 13, 15, 18 and 24 hours after morning dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: milliliter/minute (mL/min)
Arm/Group | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 16 | 16 | 16 | 17
milliliter/minute (mL/min)
  Day 1 (n=16, 16, 16, 17) | 1886 (1112) | 1434 (844.7) | 1282 (431.5) | 1440 (607.7)
  D14 (n=16, 16, 16, 16) | 1710 (1200) | 1322 (937.9) | 1292 (624.5) | 1327 (537.1)

10. Secondary Outcome: Observed Accumulation Ratio of Area Under the Curve From Time Zero to 10 Hours Postdose of PF-04991532 (Rac)
Description: Area under the curve from time zero to 10 hours postdose of PF-04991532 (AUC10) of Day 14 divided by AUC10 of Day 1
Time Frame: 0 (before morning dose), 0.5, 1, 2, 3, 4, 6, and 10 hours after morning dose on Day 1 and Day 14
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 16 | 16 | 16 | 16
ratio | 1.095 (0.3520) | 1.049 (0.2995) | 0.9004 (0.3353) | 1.017 (0.2946)

11. Secondary Outcome: Observed Accumulation Ratio of Maximum Observed Plasma Concentration of PF-04991532 After Morning Dose Administration (Rac, Cmax(AM))
Description: Maximum observed plasma concentration of PF-04991532 after morning dose administration (Cmax(AM)) of Day 14 divided by Cmax(AM) of Day 1
Time Frame: 0 (before morning dose), 0.5, 1, 2, 3, 4, 6, and 10 hours after morning dose on Day 1 and Day 14
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 16 | 16 | 16 | 16
ratio | 1.057 (0.6267) | 0.9655 (0.5913) | 0.7022 (0.4744) | 0.8663 (0.3648)

12. Secondary Outcome: Dose Normalized Area Under the Curve From Time Zero to 24 Hours Postdose (AUC24(dn)) of PF-04991532
Description: Area under the curve from time zero to 24 Hours Postdose (AUC24) divided by total daily dose
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL/mg
Arm/Group | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 16 | 16 | 16 | 17
ng*hr/mL/mg
  Day 1 (n=16, 16, 16, 17) | 4.416 (1.723) | 5.810 (2.520) | 6.497 (2.578) | 5.787 (2.540)
  Day 14 (n=16, 16, 16, 16) | 4.874 (2.271) | 6.307 (3.107) | 6.449 (2.279) | 6.275 (2.558)

13. Secondary Outcome: Dose Normalized Maximum Plasma Concentration After Morning Dose Administration (Cmax(AM)(dn)) of PF-04991532
Description: Maximum Observed Plasma Concentration of PF-04991532 after Morning Dose Administration (Cmax(AM)) divided by dose
Time Frame: 0 (before morning dose), 0.5, 1, 2, 3, 4, 6, and 10 hours after morning dose on Day 1 and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 17 | 16 | 16 | 17
ng/mL/mg
  Day 1 (n=17, 16, 16, 17) | 2.754 (1.147) | 3.245 (2.431) | 4.283 (1.947) | 3.252 (1.842)
  Day 14 (n=16, 16, 16, 16) | 2.964 (1.484) | 3.132 (3.296) | 3.009 (1.631) | 2.732 (1.530)

14. Secondary Outcome: Change From Baseline (Day -2) in Mean Daily Glucose at Day 13
Description: Mean daily glucose (MDG) was calculated based on the mean of 8 glucose measurements at pre-specified time points throughout the day.
Time Frame: Baseline: hours -72, -70, -68, -66, -62, -60, -57, and -54 on Day -2 (Day 1 morning dose was hour 0); Day 13: 0 (before morning dose), 2, 4, 6, 10, 12, 15 and 18 hours after Day 13 morning dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
mg/dL
  Baseline (Day -2) | 214.31 (42.39) | 230.70 (37.88) | 207.98 (35.10) | 219.59 (43.78) | 204.68 (45.07)
  Change from Baseline (Day 13) | 18.78 (39.66) | -27.22 (25.34) | -15.78 (31.99) | -17.29 (17.75) | -33.58 (37.06)
Statistical Analysis 1: Comparison: Placebo vs PF-04991532 25 mg; Test-to-Reference ratio and 90% confidence interval (CI) were based on adjusted geometric mean. Natural log-transformed change from baseline in MDG (Day 13) was analyzed using ANCOVA with country and treatment as fixed effect and log-transformed baseline as covariate. Placebo is the reference; the active drug group is the test; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 82.69, 90% CI 2-sided [76.06 to 89.90]
Statistical Analysis 2: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 85.39, 90% CI 2-sided [78.60 to 92.77]
Statistical Analysis 3: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 85.37, 90% CI 2-sided [78.59 to 92.76]
Statistical Analysis 4: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 75.82, 90% CI 2-sided [69.78 to 82.39]
Statistical Analysis 5: Comparison: Placebo vs PF-04991532 75 mg; Treatment difference and 90% confidence interval (CI) were based on adjusted geometric mean; Test type: Superiority or Other; Difference between Test and Reference = -35.84, 90% CI 2-sided [-52.89 to -18.78]

15. Secondary Outcome: Change From Baseline in Area Under the Curve of Glucose From Time 2 to 6 Hours Post Morning Dose (Glucose AUC(2-6)) Following Mixed Meal Tolerance Test (MMTT) at Day 14
Description: Area under the curve of glucose from time 2 to 6 hours post morning dose (Glucose AUC(2-6)) was calculated based on 8 glucose measurements at prespecified time points using the linear trapezoidal method. Nominal times were used in the calculation. Liquid meal was administered 2 hours post morning dose of PF-04991532 for mixed meal tolerance test (MMTT).
Time Frame: Baseline: hours -46, -45.75, -45.5, -45, -44.5, -44, -43, -and -42 on Day -1 (Day 1 morning dose was hour 0); Day 14: 2, 2.25, 2.5, 3, 3.5, 4, 5, and 6 hours after Day 14 morning dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
mg*hr/dL
  Baseline (Day -1) | 1091.23 (163.30) | 1126.34 (119.26) | 1029.76 (154.84) | 1085.84 (245.64) | 1050.69 (241.70)
  Change from Baseline (Day 14) | 86.05 (148.94) | -84.44 (99.91) | -12.65 (114.19) | -60.55 (89.36) | -158.93 (152.09)
Statistical Analysis 1: Comparison: Placebo vs PF-04991532 25 mg; Test-to-Reference ratio and 90% confidence interval (CI) were based on adjusted geometric mean. Natural log-transformed change from baseline in Glucose AUC(2-6) was analyzed using ANCOVA with country and treatment as fixed effect and log-transformed baseline as covariate. Placebo is the reference; the active drug group is the test; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 86.72, 90% CI 2-sided [81.13 to 92.70]
Statistical Analysis 2: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 91.13, 90% CI 2-sided [85.24 to 97.44]
Statistical Analysis 3: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 87.05, 90% CI 2-sided [81.44 to 93.04]
Statistical Analysis 4: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 77.95, 90% CI 2-sided [72.91 to 83.34]

16. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: The average of the Day -1 (hour -48), Day 0 (hour -24) and Day 1 pre-dose (hour 0) measurements was the baseline for fasting plasma glucose (FPG) analyses.
Time Frame: Baseline: hour -48 on Day -1, hour -24 on Day 0, and hour 0 (before morning dose) on Day 1; hour 0 (before morning dose of each day) on Days 1, 2, 3, 6, and 10; and 24 hours after Day 14 morning dose on Day 15
Population: The pharmacodynamic analysis population was defined as all randomized participants who received at least 1 dose of study medication (PF-04991532 or placebo) and had at least 1 of the pharmacodynamic parameters of interest; "n" is the number of participants analyzed for each day.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 16 | 17 | 16 | 16 | 17
mg/dL
  Day 2 (n=16, 17, 16, 16, 17) | -4.19 (17.77) | -5.04 (10.43) | -4.33 (18.15) | 0.29 (14.93) | -5.55 (36.08)
  Day 3 (n=16, 17, 16, 16, 17) | -0.63 (15.76) | -8.92 (11.86) | -2.15 (15.25) | 0.23 (14.06) | -7.78 (16.40)
  Day 6 (n=16, 16, 16, 16, 16) | 3.44 (26.69) | -9.40 (16.68) | -9.90 (18.13) | -6.33 (12.24) | -16.90 (23.67)
  Day 10 (n=16, 16, 16, 16, 16) | -10.88 (43.97) | -17.21 (24.08) | -16.96 (26.78) | -10.33 (15.75) | -17.40 (30.99)
  Day 14 (n=16, 16, 16, 16, 16) | 9.00 (26.90) | -17.83 (25.71) | -14.52 (23.08) | -7.27 (8.78) | -11.40 (19.12)
  Day 15 (n=16, 16, 16, 16, 15) | 12.63 (44.47) | -9.71 (25.96) | -8.15 (22.81) | -0.58 (16.71) | -4.22 (37.34)
Statistical Analysis 1: Comparison: Placebo vs PF-04991532 25 mg; Test-to-Reference ratio of log-transformed change from baseline and 90% confidence interval (CI) of log-transformed change from baseline at Day 2 were based on adjusted geometric mean. Natural log-transformed change from baseline in FPG was analyzed using mixed effects model with country, treatment as fixed effect and log-transformed baseline as covariate. Placebo is the reference; the active drug group is the test; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 2 = 100.04, 90% CI 2-sided [92.70 to 107.96]
Statistical Analysis 2: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 2 = 99.44, 90% CI 2-sided [92.04 to 107.43]
Statistical Analysis 3: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 2 = 101.67, 90% CI 2-sided [94.10 to 109.84]
Statistical Analysis 4: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 2 = 96.82, 90% CI 2-sided [89.69 to 104.52]
Statistical Analysis 5: Comparison: Placebo vs PF-04991532 25 mg; Test-to-Reference ratio of log-transformed change from baseline and 90% confidence interval (CI) of log-transformed change from baseline at Day 3 were based on adjusted geometric mean. Natural log-transformed change from baseline in FPG was analyzed using mixed effects model with country, treatment as fixed effect and log-transformed baseline as covariate. Placebo is the reference; the active drug group is the test; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 3 = 95.85, 90% CI 2-sided [88.82 to 103.44]
Statistical Analysis 6: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 16, analysis 5]; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 3 = 98.71, 90% CI 2-sided [91.37 to 106.64]
Statistical Analysis 7: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 16, analysis 5]; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 3 = 99.72, 90% CI 2-sided [92.30 to 107.73]
Statistical Analysis 8: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 16, analysis 5]; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 3 = 94.49, 90% CI 2-sided [87.53 to 102.10]
Statistical Analysis 9: Comparison: Placebo vs PF-04991532 25 mg; Test-to-Reference ratio of log-transformed change from baseline and 90% confidence interval (CI) of log-transformed change from baseline at Day 6 were based on adjusted geometric mean. Natural log-transformed change from baseline in FPG was analyzed using mixed effects model with country, treatment as fixed effect and log-transformed baseline as covariate. Placebo is the reference; the active drug group is the test; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 6 = 93.43, 90% CI 2-sided [86.50 to 100.91]
Statistical Analysis 10: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 16, analysis 9]; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 6 = 92.71, 90% CI 2-sided [85.81 to 100.15]
Statistical Analysis 11: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 16, analysis 9]; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 6 = 94.08, 90% CI 2-sided [87.08 to 101.64]
Statistical Analysis 12: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 16, analysis 9]; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 6 = 87.74, 90% CI 2-sided [81.20 to 94.81]
Statistical Analysis 13: Comparison: Placebo vs PF-04991532 25 mg; Test-to-Reference ratio of log-transformed change from baseline and 90% confidence interval (CI) of log-transformed change from baseline at Day 10 were based on adjusted geometric mean. Natural log-transformed change from baseline in FPG was analyzed using mixed effects model with country, treatment as fixed effect and log-transformed baseline as covariate. Placebo is the reference; the active drug group is the test; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 10 = 96.91, 90% CI 2-sided [89.72 to 104.67]
Statistical Analysis 14: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 10 = 96.05, 90% CI 2-sided [88.90 to 103.76]
Statistical Analysis 15: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 10 = 99.63, 90% CI 2-sided [92.21 to 107.64]
Statistical Analysis 16: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 10 = 94.50, 90% CI 2-sided [87.46 to 102.11]
Statistical Analysis 17: Comparison: Placebo vs PF-04991532 25 mg; Test-to-Reference ratio of log-transformed change from baseline and 90% confidence interval (CI) of log-transformed change from baseline at Day 14 were based on adjusted geometric mean. Natural log-transformed change from baseline in FPG was analyzed using mixed effects model with country, treatment as fixed effect and log-transformed baseline as covariate. Placebo is the reference; the active drug group is the test; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 14 = 86.75, 90% CI 2-sided [80.32 to 93.69]
Statistical Analysis 18: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 16, analysis 17]; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 14 = 87.87, 90% CI 2-sided [81.34 to 94.93]
Statistical Analysis 19: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 16, analysis 17]; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 14 = 91.35, 90% CI 2-sided [84.55 to 98.70]
Statistical Analysis 20: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 16, analysis 17]; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 14 = 88.60, 90% CI 2-sided [82.00 to 95.74]
Statistical Analysis 21: Comparison: Placebo vs PF-04991532 25 mg; Test-to-Reference ratio of log-transformed change from baseline and 90% confidence interval (CI) of log-transformed change from baseline at Day 15 were based on adjusted geometric mean. Natural log-transformed change from baseline in FPG was analyzed using mixed effects model with country, treatment as fixed effect and log-transformed baseline as covariate. Placebo is the reference; the active drug group is the test; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 15 = 90.45, 90% CI 2-sided [83.75 to 97.69]
Statistical Analysis 22: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 16, analysis 21]; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 15 = 90.45, 90% CI 2-sided [84.03 to 98.08]
Statistical Analysis 23: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 16, analysis 21]; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 15 = 94.75, 90% CI 2-sided [87.69 to 102.34]
Statistical Analysis 24: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 16, analysis 21]; Test type: Superiority or Other; Test-to-Reference Ratio (%) at Day 15 = 93.18, 90% CI 2-sided [86.17 to 100.77]

17. Secondary Outcome: Change From Baseline in Area Under the Curve of Insulin From Time 2 to 6 Hours Post Morning Dose (Insulin AUC(2-6)) Following Mixed Meal Tolerance Test (MMTT) at Day 14
Description: Area Under the Curve of Insulin from Time 2 to 6 Hours Post Morning Dose (Insulin AUC(2-6)) was calculated based on 8 insulin measurements at prespecified time points using the linear trapezoidal method. Nominal times were used in the calculation. Liquid meal was administered 2 hours post morning dose of PF-04991532 for mixed meal tolerance test (MMTT).
Time Frame: as for outcome 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliUnit*hour/liter (mU*hr/L)
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 16 | 13 | 15 | 14 | 14
milliUnit*hour/liter (mU*hr/L)
  Baseline (Day -1) | 149.12 (117.08) | 139.40 (77.81) | 166.87 (132.39) | 111.13 (69.16) | 276.61 (313.03)
  Change from Baseline (Day 14) | -3.96 (18.09) | 15.87 (27.16) | -3.06 (32.79) | 11.82 (24.87) | -38.06 (73.89)
Statistical Analysis 1: Comparison: Placebo vs PF-04991532 25 mg; Test-to-Reference ratio and 90% confidence interval (CI) were based on adjusted geometric mean. Natural log-transformed change from baseline in Insulin AUC(2-6) (Day 14) was analyzed using ANCOVA with country and treatment as fixed effect and log-transformed baseline as covariate. Placebo is the reference; the active drug group is the test; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 112.83, 90% CI 2-sided [99.84 to 127.50]
Statistical Analysis 2: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 102.11, 90% CI 2-sided [90.78 to 114.85]
Statistical Analysis 3: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 111.04, 90% CI 2-sided [98.50 to 125.18]
Statistical Analysis 4: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 96.73, 90% CI 2-sided [85.46 to 109.48]

18. Secondary Outcome: Change From Baseline in Area Under the Curve of C-peptide From Time 2 to 6 Hours Post Morning Dose (C-peptide AUC(2-6)) Following Mixed Meal Tolerance Test (MMTT) at Day 14
Description: Area Under the Curve of C-peptide from Time 2 to 6 Hours Post Morning Dose (C-peptide AUC(2-6)) was calculated based on 8 C-peptide measurements at prespecified timepoints using the linear trapezoidal method. Nominal times were used in the calculation. Liquid meal was administered 2 hours post morning dose of PF-04991532 for mixed meal tolerance test (MMTT).
Time Frame: as for outcome 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
ng*hr/mL
  Baseline (Day -1) | 15.79 (6.08) | 17.04 (6.73) | 17.20 (5.89) | 15.23 (4.51) | 19.21 (7.61)
  Change from Baseline (Day 14) | 0.09 (2.15) | 1.34 (2.64) | -1.53 (2.88) | -0.55 (1.63) | -2.12 (2.97)
Statistical Analysis 1: Comparison: Placebo vs PF-04991532 25 mg; Test-to-Reference ratio and 90% confidence interval (CI) were based on adjusted geometric mean. Natural log-transformed change from baseline in C-peptide AUC(2-6) (Day 14) was analyzed using ANCOVA with country and treatment as fixed effect and log-transformed baseline as covariate. Placebo is the reference; the active drug group is the test; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 107.13, 90% CI 2-sided [98.69 to 116.30]
Statistical Analysis 2: Comparison: Placebo vs PF-04991532 75 mg; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 92.57, 90% CI 2-sided [85.26 to 100.50]
Statistical Analysis 3: Comparison: Placebo vs PF-04991532 150 mg; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 96.07, 90% CI 2-sided [88.51 to 104.27]
Statistical Analysis 4: Comparison: Placebo vs PF-04991532 300 mg; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; Test-to-Reference Ratio (%) = 91.70, 90% CI 2-sided [84.38 to 99.65]

19. Secondary Outcome: Change From Baseline in Fasting Lipid Parameters at Day 14 and 16
Description: Baseline for fasting triglycerides (TG) was defined as the average of the Day -1 (hour -48), Day 0 (hour -24), and Day 1 pre-dose (hour 0) measurements. Baseline for fasting total cholesterol (TC), cholesterol (high-density lipoprotein (HDL)), and cholesterol (low-density lipoprotein (LDL)) was defined as the Day 1 pre-dose (hour 0) measurement.
Time Frame: Baseline: hour -48 on Day -1, hour -24 on Day 0, and hour 0 on Day 1 for TG and Hour 0 (before morning dose) on Day 1 for TC, HDL, and LDL; 48 hours after morning dose on Day 16 for TG and Hour 0 (before morning dose) on Day14 for TC, HDL, and LDL
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
mg/dL
  Triglycerides (Day 16) (n=16, 16, 16, 16, 16) | -9.81 (35.87) | 12.79 (45.64) | 37.52 (98.13) | 18.24 (36.08) | 58.00 (67.31)
  Total Cholesterol (Day 14) (n=16, 16, 16, 15, 16) | 0.06 (16.98) | -11.75 (31.62) | 4.19 (20.04) | 1.80 (19.29) | 11.38 (30.17)
  Cholesterol HDL (Day 14) (n=16, 16, 16, 16, 16) | 1.75 (4.48) | -1.88 (7.75) | 1.88 (6.04) | 0.69 (8.44) | 3.94 (7.17)
  Cholesterol LDL (Day 14) (n=16, 16, 15, 14, 15) | 2.38 (17.64) | -8.06 (26.98) | 4.67 (22.48) | -0.79 (16.40) | 1.53 (25.53)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | PF-04991532 25 mg | PF-04991532 75 mg | PF-04991532 150 mg | PF-04991532 300 mg
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 0/16 | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 4/16 | 3/17 | 7/16 | 5/16 | 4/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | PF-04991532 25 mg (N=17) | PF-04991532 75 mg (N=16) | PF-04991532 150 mg (N=16) | PF-04991532 300 mg (N=17)
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Infusion site swelling (General disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Carbuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 1 | 0 | 0
Electrocardiogram ST-T change (Investigations) | 0 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 3 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.